CLINICAL TRIAL: NCT05682391
Title: The Impact of Postoperative Bed Rest on the Repair of Cerebrospinal Fluid (CSF) Leakage After Transnasal Transsphenoidal Pituitary Surgery
Brief Title: Bed Rest on the Effect of CSF Leakage Repair After Transsphenoidal Pituitary Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202207083RINA
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Adenoma Pituitary; CSF Leakage
Keywords: CSF leakage; transsphenoidal adenomectomy; bed rest
MeSH Terms: conditions — Pituitary Neoplasms; Cerebrospinal Fluid Rhinorrhea | interventions — Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Prospective experimental - no bed rest after intraoperative leak (No Intervention): Randomized after surgery if intraoperative CSF leakage occurs. The ratio for allocating into arm 1 vs. arm 2 is 2:1.
- Prospective control - bed rest after intraoperative leak (Active Comparator): Randomized after surgery if intraoperative CSF leakage occurs. The ratio for allocating into arm 1 vs. arm 2 is 2:1.
  Interventions: Other: Bed rest
- Prospective control - no bed rest after no intraoperative leak (No Intervention): Enters this arm if no intraoperative CSF leakage occurs.
- Retrospective control - bed rest after intraoperative leak (Active Comparator): Historical control, bed rest applied after intraoperative CSF leakage.
  Interventions: Other: Bed rest
- Retrospective control - no bed rest after no intraoperative leak (No Intervention): Historical control, bed rest not applied after no intraoperative CSF leakage.

INTERVENTIONS:
Other: Bed rest — Strict bed rest ordered after surgery that does not allow the participant to elevate the head of bed over 30 degrees
  Arms: Prospective control - bed rest after intraoperative leak; Retrospective control - bed rest after intraoperative leak

SUMMARY:
Postoperative cerebrospinal fluid (CSF) leakage is a well-known complication that might occur after transnasal transsphenoidal adenomectomy at an incidence of 0.5-15% according to different literature reports. Persistent CSF leakage may lead to intracranial hypotension or meningitis, therefore aggressive management is mandatory. The treatment is immediate repair during transsphenoidal surgery once intraoperative CSF leakage is identified, with the adjunct of postoperative bed rest and/or lumbar drainage. However, due to the advances in endoscopic endonasal skull base surgery, some surgical teams have advocated that postoperative bed rest may not be necessary if appropriate repair have been performed. High-flow CSF leakage typically occurs in an extended endonasal approach to the anterior or posterior cranial fossa, whereas CSF leakage resulting from transsphenoidal pituitary surgery is usually easier to be repaired.

Bed rest is stressful management for patients and poses increased risks in many ways, such as the need for an indwelling urinary catheter, musculoskeletal pain, affected sleep quality, and increased possibility of thromboembolism. It is crucial that the duration of bed rest be cut short or totally avoided if clinically acceptable. In reviewing the literature, there is insufficient evidence supporting the routine use of postoperative bed rest after CSF leakage repair in transsphenoidal surgery. This study aims to compare the efficacy of successful CSF leakage repair with or without postoperative bed rest with an open-label randomized trial design.

DETAILED DESCRIPTION:
Postoperative CSF leakage is a well-known complication that might occur after transnasal transsphenoidal adenomectomy at an incidence of 0.5-15% according to different literature reports. Persistent CSF leakage may lead to intracranial hypotension or meningitis, therefore aggressive management is mandatory. The reason that a postoperative CSF leakage would occur mostly is due to the rupture of arachnoid membrane caused by intraoperative manipulation, resulting in direct communication between the subarachnoid space and the nasal cavity. Even when in cases without intraoperative CSF leakage detected, there is a reported incidence of 1.3% of postoperative CSF leakage.

The rate of intraoperative CSF leakage varies in different tumor sizes, tumor extents, tumor natures, and surgical teams, and it could not be precisely documented as 23.3-60% were reported. The treatment is immediate repair during transsphenoidal surgery once intraoperative CSF leakage is identified, with the adjunct of postoperative bed rest and/or lumbar drainage. However, due to the advances in endoscopic endonasal skull base surgery, some surgical teams have advocated that postoperative bed rest may not be necessary if appropriate repair have been performed. High-flow CSF leakage typically occurs in an extended endonasal approach to the anterior or posterior cranial fossa, whereas CSF leakage resulting from transsphenoidal pituitary surgery is usually easier to be repaired.

Bed rest is stressful management for patients and poses increased risks in many ways, such as the need for an indwelling urinary catheter, musculoskeletal pain, affected sleep quality, and increased possibility of thromboembolism. It is crucial that the duration of bed rest be cut short or totally avoided if clinically acceptable. In reviewing the literature, there is insufficient evidence supporting the routine use of postoperative bed rest after CSF leakage repair in transsphenoidal surgery. This study aims to compare the efficacy of successful CSF leakage repair with or without postoperative bed rest with an open-label randomized trial design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pituitary adenoma requiring surgical resection.

Exclusion Criteria:

* Spontaneous CSF leakage occurs prior to transsphenoidal surgery.
* The growth of adenoma extends to anterior cranial fossa or clival region.
* The growth of adenoma extends to 3rd ventricle.
* Prior history of transsphenoidal surgery.
* Prior history of radiotherapy or radiosurgery to the sella or nearby skull base region.
* Class 2 obesity or extremely obese: BMI ≧35.
* Pregnant or lactating women.
* Patients who could not give informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of CSF leakage within 3 months postoperatively | 12 weeks after the date of surgery
  Any documented CSF leakage within 3 months postoperatively. Confirmation of CSF leakage could either be:
  1. typical symptoms of CSF rhinorrhea, plus visible clear and colorless rhinorrhea with positive glucose response
  2. atypical symptoms of CSF rhinorrhea, plus visualization of clear and colorless fluid from the operative site via sinoscope
  3. atypical symptoms of CSF rhinorrhea, plus identifiable fluid accumulation in the sphenoid sinus and suspicious site of CSF fistula via neuroimaging modalities

SECONDARY OUTCOMES:
Occurrence of meningitis within 3 months postoperatively | 12 weeks after the date of surgery
  Any documented meningitis within 3 months postoperatively.
Length of hospital stay | 24 weeks after the date of surgery
  The length of stay is calculated from 1 day prior to surgery until the day of discharge.
Results of 36-Item short form health survey (SF-36) surveys | On postoperative day 1, postoperative day 7, postoperative day 28, postoperative week 12 and postoperative week 24.
  SF-36 with its 8 subscales as well as the physical component summary (PCS) and mental component summary (MCS) scores. Each of the 8 subscales (physical functioning [PF], role physical [RP], bodily pain [BP], general health [GH], vitality [VT], social functioning [SF], role emotional [RE], and mental health [MH]) has a minimum value of 0 and maximum value of 100, a higher score relates to a better outcome. The PCS score is the average score of PF, RP, BP, and GH, while the MCS score is the average score of VT, SF, RE, and MH (both has the minimum value of 0 and maximum value of 100, a higher score relates to a better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neurosurgery, Department of Surgery, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No